CLINICAL TRIAL: NCT05971498
Title: Assessment of Anxiety, Depression, Sleep Quality and Quality of Life in Systemic Lupus Erythematosus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, Principal investigator, Assiut University
Other Study IDs: AssiutU SLE
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- cases
- control

SUMMARY:
The goal of this case control observational study is to asses anxiety, sleep, depression and quality of life in Systemic Lupus Erythematosus (SLE) patients.

The main aims are:

* asses anxiety, sleep, depression and quality of life in SLE patients
* their relation to disease activity

we will compare SLE patients to healthy subjects.

DETAILED DESCRIPTION:
All patients will be subjected to clinical evaluation (full history and examination, laboratory evaluation (include erythrocyte sedimentation rate (ESR) measured by standard westergren method (mm/h), serum C-reactive protein (CRP), complete blood count (CBC), serum urea and creatinine, aspartate transaminase (AST), alanine transaminase (ALT), complete urine analysis for: urinary casts (hyaline, granular), hematuria (RBCs/ high power field), pyuria (WBCs/ high power field), 24-hour urinary protein and creatinine clearance. Immunological work up will include antinuclear antibodies (ANA) by ELISA, anti-double stranded DNA (ds-DNA) by ELISA and complement components C3 and C4 by nephelometry. Disease activity will be assessed via SLE disease activity index (SLEDAI): SLEDAI is based on the presence of 24 descriptors in nine organ systems over the preceding 30 days. Descriptors of SLEDAI are documented as present or absent. Each of the descriptors has a weighted score and the total score of SLEDAI is the sum of all 24 descriptor scores. The total score falls between 0 and 105, with higher scores representing higher disease activity.

Psychological assessment will be performed according to the following scales

* Hamilton Anxiety Rating Scale (HAM-A): It consists of 14 items and measures both psychic and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where a score ≤ 17 indicates mild anxiety, 18-24 mild to moderate anxiety, , 25-30 moderate to severe anxiety and scores >30 indicate severe anxiety.
* Hamilton Depression Rating Scale: the original scale has 21 items, but scoring is based only on the first 17. Scores less than or equal to 7 indicates normal response, 8-13 mild depression, 14-18 Moderate, 19-22 severe, and > 22 very severe depression.

Sleep quality assessment was done via

* Insomnia severity index (ISI) : contains seven domains assessing sleep-onset difficulties, sleep maintenance, sleep satisfaction, effect on daily functioning, impairment attributed to sleep problems, and distress associated with insomnia. Each item is rated on a 0-4 scale, and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
* Epworth sleepiness scale : subjects describe how often they fall asleep in certain situations on a scale of 0-3, with total scores ranging from 0 to 24. An ESS score ≥ 10 is indicative of subjective excessive daytime sleepiness and score > 16 indicates high level of daytime sleepiness.

Pittsburgh Sleep Quality Index the first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components (sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use). The scores for each component are summed to get a total score (range 0-21). A score > 5 suggests poor sleep quality.

Assessment of Health status and quality of life via short form health survey (SF36):Thirty-five of the 36 items are grouped into eight scales: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. One item assesses perception of changes in health over the last year but is not used calculate scale scores. Higher scores indicate high quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SLE according to the 2012 systemic lupus international collaborating clinics (SLICC) criteria .

Exclusion Criteria:

* Evidence of end-organ failures such as heart failure, liver cell or renal failure,
* History of psychological disorders .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SLE patients and healthy control
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of insomnia in SLE patients by Insomnia severity index | 3 MONTHS
  insomnia severity index contains seven domains assessing sleep-onset difficulties, sleep maintenance, sleep satisfaction, effect on daily functioning, impairment attributed to sleep problems, and distress associated with insomnia. Each item is rated on a 0-4 scale, and th e total score ranges from 0 to 28. A higher score suggests more severe insomnia
evaluation of excessive daytime sleepiness in SLE patients by Epworth sleepiness scale | 3 months
  Subjects describe how often they fall asleep in certain situations on a scale of 0-3, with total scores ranging from 0 to 24. An ESS score ≥ 10 is indicative of subjective excessive daytime sleepiness and score > 16 indicates high level of daytime sleepiness
evaluation of anxiety in SLE patients by hamilton anxiety rating scale | 3 months
  It consists of 14 items and measures both psychic and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where a score ≤ 17 indicates mild anxiety, 18-24 mild to moderate anxiety, , 25-30 moderate to severe anxiety and scores >30 indicate severe anxiety
evaluation of depression in SLE patients by hamilton depression rating scale | 3 months
  The original scale has 21 items, but scoring is based only on the first 17 with total score ranges from 0 to 52. Scores less than or equal to 7 indicates normal response, 8-13 mild depression, 14-18 Moderate, 19-22 severe, and > 22 very severe depression.
evaluation of QoL in SLE patients by short form health survey (sf36 ) | 3 months
  Thirty-five of the 36 items are grouped into eight scales: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. One item assesses perception of changes in health over the last year but is not used calculate scale scores. Mean score ranges from 0 to100. High scores indicate lower disability
evaluation of sleep quality and disturbances in SLE patients by Pittsburgh Sleep Quality Index | 3 months
  The first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components (sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use). The scores for each component are summed to get a total score (range 0-21). A score > 5 suggests poor sleep quality

SECONDARY OUTCOMES:
Correlation of disease activity (SLEDAI) with Hamilton anxiety rating scale, Hamilton depression rating scale, Epworth sleepiness scale,Pittsburgh Sleep Quality Index and short form health survey sf 36 | 3 months
  The SLEDAI consists of 24 items (nine organ systems) that are scored based on presence at the time of visit or in the preceding 10 days. The scoring is additive across items, with a possible total score range of 0 to 105 (higher scores represent greater disease activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut university hospital, Asyut, Egypt